CLINICAL TRIAL: NCT01829477
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, 24-Week Study to Evaluate the Efficacy and Safety of Daily Oral TAK-875 50 mg Compared With Placebo as an Add-on to Glimepiride in Subjects With Type 2 Diabetes
Brief Title: Comparison of TAK-875 to Placebo as an Add-on to Glimepiride in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to potential concerns about liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_309; 2013-000007-17 (EudraCT Number); U1111-1138-8680 (Registry Identifier: WHO); 164539 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAK-875 50 mg (Experimental): TAK-875 50 mg tablet, orally, once daily and glimepiride 6 mg (or Maximum Tolerated Dose), tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: TAK-875; Drug: Glimepiride
- Placebo (Placebo Comparator): TAK-875 placebo-matching tablet, orally, once daily and glimepiride 6 mg (or Maximum Tolerated Dose), tablets, orally, once daily for up to 24 weeks.
  Interventions: Drug: TAK-875 Placebo; Drug: Glimepiride

INTERVENTIONS:
Drug: TAK-875 — TAK-875 50 mg tablets
  Arms: TAK-875 50 mg
Drug: TAK-875 Placebo — TAK-875 placebo-matching tablets
  Arms: Placebo
Drug: Glimepiride — Glimepiride tablet.
  Other Names: Amaryl

SUMMARY:
The purpose of this study is to evaluate the effect of TAK-875 compared to placebo on glycemic control over a 24-week Treatment Period when used as an add-on to glimepiride in addition to diet and exercise.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-875. TAK-875 is being tested to treat people who have diabetes. This study will look at glycosylated hemoglobin (blood glucose combined with hemoglobin, also known as HbA1c) and blood sugar levels in people who take TAK-875 in addition to glimepiride and diet and exercise.

The study will enroll approximately 260 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-875 50 mg
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take one tablet at the same time each day throughout the study. This multi-center trial will be conducted in North America and Europe. The overall time to participate in this study is up to 44 weeks and participants will make up to 17 visits to the clinic.

Due to potential concerns about liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Male or female and aged 18 or older with a historical diagnosis of type 2 diabetes mellitus (T2DM).
4. Has a glycosylated hemoglobin (HbA1c) of 7.0% to10.0%, inclusive at screening, and has been treated with diet and exercise and a sulfonylurea for at least 12 weeks.
5. Has a body mass index (BMI) ≤45 kg/m2 at Screening.
6. Participants regularly using other, non-excluded medications, must be on a stable dose and regimen for at least 4 weeks prior to Screening. However, as needed (PRN) use of prescription or over-the-counter medication is allowed at the discretion of the investigator. Note: Participants who require initiation of a chronically administered medication(s) due to a disease or condition diagnosed at Screening must be re-screened after the new regimen has been stabilized.
7. A female of childbearing potential who is sexually active with a non-sterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose of study drug.
8. Is able and willing to monitor glucose with a sponsor-provided home glucose monitor and consistently record his or her own blood glucose concentrations and participant diaries.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening or has received an investigational antidiabetic drug within 3 months prior to Screening.
2. Has participated in a previous TAK-875 study.
3. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
5. Has a hemoglobin ≤12 g/dL (≤120 gm/L) for males and ≤10 g/dL (≤100 gm/L) for females at Screening.
6. Has a systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥95 mm Hg at Screening (If the participant meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after the initial measurement and decision will be made based on the second measurement).
7. Has a history of cancer that has been in remission for <5 years prior to Screening. A history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed.
8. Has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2.0x the upper limit of normal (ULN) at Screening.
9. Has a total bilirubin level greater than the ULN at Screening. Exception: if a participant has documented Gilbert's Syndrome, the participant will be allowed with an elevated bilirubin level per the investigator's discretion.
10. Has a serum creatinine ≥1.5 mg/dL (≥133 μmol/L) [if male] or ≥1.4 mg/dL (≥124 μmol/L) [if female] and/or estimated (based on Modification of Diet in Renal Disease [MDRD] calculation) glomerular filtration rate (GFR) <60 mL/min/1.73m2 (regardless of gender) at Screening.
11. Has uncontrolled thyroid disease.
12. Has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
13. Has had gastric banding or gastric bypass surgery within 1 year prior to Screening.
14. Has known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency, which increases risk for hemolytic anemia by sulfonylurea treatment.
15. Has a known history of infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
16. Had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram (ECG), cerebrovascular accident or transient ischemic attack within 3 months prior or at Screening.
17. Has a history of hypersensitivity, allergies, or has had an anaphylactic reaction(s) to any component of TAK-875 or glimepiride.
18. Has a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse within 2 years prior to Screening.
19. Received excluded medications prior to Screening or is expected to receive excluded medication.
20. If female, the participant is pregnant (confirmed by laboratory testing, ie, serum human chorionic gonadotropin (hCG), in females of childbearing potential) or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
21. Is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent is available.
22. Has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the participant according to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (69):
- United States (38):
  - Muscle Shoals, Alabama
  - Phoenix, Arizona
  - Fresno, California
  - Long Beach, California
  - National City, California
  - North Hollywood, California
  - Pismo Beach, California
  - Lakewood, Colorado
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Coral Gables, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Conyers, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Oxon Hill, Maryland
  - Flint, Michigan
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Haddon Heights, New Jersey
  - Rosedale, New York
  - Morehead City, North Carolina
  - Morganton, North Carolina
  - Maumee, Ohio
  - Hanleysville, Pennsylvania
  - Uniontown, Pennsylvania
  - Laurens, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Tomball, Texas
  - Manassas, Virginia
- Bulgaria (3):
  - Gabrovo
  - Plovdiv
  - Sofia
- Canada (3):
  - Oakville, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
- Hungary (5):
  - Budapest
  - Gödöllő
  - Kistelek
  - Komárom
  - Zalaegerszeg
- Poland (10):
  - Bialystok
  - Gdansk
  - Grodzisk Mazowiecki
  - Kamieniec Ząbkowicki
  - Lodz
  - Oświęcim
  - Poznan
  - Puławy
  - Rzeszów
  - Zgierz
- Romania (3):
  - Baia Mare
  - Ploieşti
  - Timișoara
- Slovakia (7):
  - Banská Bystrica
  - Bratislava
  - Dolný Kubín
  - Levice
  - Lučenec
  - Pezinok
  - Svidník

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in the United States, Slovakia, Bulgaria, Hungary, and Canada from 19 April 2013 to 11 February 2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus (T2DM), inadequately controlled when treated with only diet, exercise and a sulfonylurea for at least 12 weeks prior to screening, were enrolled in 1 of 2 treatment groups: placebo; fasiglifam 50 milligram (mg).
Groups:
- Placebo: Fasiglifam placebo-matching tablet, orally, once daily and glimepiride 6 mg (or maximum tolerated dose), tablet, orally, once daily for up to 24 weeks.
- Fasiglifam 50 mg: Fasiglifam 50 mg, tablet, orally, once daily and glimepiride 6 mg (or maximum tolerated dose), tablet, orally, once daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Fasiglifam 50 mg
Started | 17 | 16
Completed | 1 | 1
Not Completed | 16 | 15
Not completed — Study Terminated by Sponsor | 15 | 15
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fasiglifam 50 mg | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Customized [Number; unit: Participants]
  18 to 64 years | 10 (11.82) | 12 (9.70) | 22
  65 to 84 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 1 | 4
  White | 14 | 15 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 5 | 2 | 7
  Not Applicable | 6 | 9 | 15
Baseline Glycosylated Hemoglobin (HbA1c) Category [Number; unit: participants]
  Less Than (<) 8.5 Percent (%) | 10 | 11 | 21
  Greater Than or Equal to (>=) 8.5% | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 relative to baseline.
Time Frame: Baseline and Week 24
Population: In accordance with the Statistical Analysis Plan (SAP), due to the limited enrollment at the time of study termination, the summaries and statistical analyses of primary and secondary efficacy parameters originally intended and described in the protocol were not produced.
Arm/Group | Placebo | Fasiglifam 50 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With HbA1c <7 % at Week 24.
Time Frame: Week 24
Population: In accordance with the SAP, due to the limited enrollment at the time of study termination, the summaries and statistical analyses of primary and secondary efficacy parameters originally intended and described in the protocol were not produced.
Arm/Group | Placebo | Fasiglifam 50 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: The change between the fasting plasma glucose value collected at week 24 or final visit relative to baseline.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Arm/Group | Placebo | Fasiglifam 50 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after the last dose of double-blinded study drug.
Description: At each visit, the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Fasiglifam 50 mg
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 5/17 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Fasiglifam 50 mg (N=16)
Hypoesthesia (Nervous system disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Electrocardiogram (ECG) abnormal (Investigations) | 0 | 1
Episcleritis (Eye disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.